CLINICAL TRIAL: NCT02027155
Title: A Phase I, Randomized, Double-blind, Placebo-controlled, Rising-dose Study to Assess the Tolerability, Safety, Pharmacokinetics, and Pharmacodynamics of Single IV Doses of AR09 in Healthy Subjects
Brief Title: Phase I Rising-dose Study to Assess Tolerability, Safety, Pharmacokinetics, Pharmacodynamics of AR09
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study stopping criteria was met
Sponsor: Arbor Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Other
Other Study IDs: AR09.001; AR09.001 (Other: IND)
Record Dates: First submitted 2013-12-29; First posted 2014-01-06 (Estimated); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Anesthesia
Keywords: healthy volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AR09 solution (Active Comparator): AR09, Randomized, Double-blind, Placebo-controlled, Rising-dose Study to Assess the Tolerability, Safety, Pharmacokinetics, and Pharmacodynamics of Single IV Doses of AR09 in Healthy Subjects
  Interventions: Drug: AR09 solution; Drug: placebo
- Placebo (for AR09 solution) (Placebo Comparator): Placebo; normal saline
  Interventions: Drug: AR09 solution; Drug: placebo

INTERVENTIONS:
Drug: AR09 solution — moderate levels of sedation
  Other Names: investigational product
Drug: placebo — Sterile Saline, USP
  Other Names: Sterile Saline, United States Pharmacopeial (USP)

SUMMARY:
This will be a randomized, double-blind, placebo-controlled, rising-dose study of single IV doses of AR09 in healthy subjects. Each infusion will occur over 10 minutes.

DETAILED DESCRIPTION:
Each subject will complete Screening, Baseline, Treatment, and Follow-Up Phases. The Screening Phase will be conducted on an outpatient basis within 30 days, but no less than 3 days, prior to the start of the Baseline Phase. The Baseline Phase will consist of clinical research unit (CRU) admission and final qualification assessments. The Treatment Phase will be comprised of dosing on Day 1, post-treatment safety and pharmacodynamic assessments, and blood and urine collection. Subjects may be discharged approximately 24 hours after study drug administration on Day 2, provided the Modified Aldrete Score and all designated discharge criteria are clinically acceptable to the Investigator. The Follow-Up Phase will occur on Study Day 5 (± 1 day).

ELIGIBILITY:
Inclusion Criteria:

* Males/females between 18 to 50 years of age, inclusive;
* Body mass index 18 to 30 kg/m2, inclusive.
* All females must have a negative serum beta human chorionic gonadotropin test result at screening and a negative urine pregnancy test result at baseline. Female subjects must be either post-menopausal, surgically sterile or using an acceptable method of contraception. Acceptable surgical sterilization techniques are hysterectomy, bilateral tubal ligation with surgery at least 6 months prior to dosing and bilateral oophorectomy with surgery at least 2 months prior to dosing. Acceptable methods of contraception are an intrauterine device, contraceptive implant, oral contraceptive (stable dose of the same hormonal contraceptive product for at least 12 weeks prior to dosing), a vasectomized partner and a double-barrier method (condom + spermicide / diaphragm + spermicide).
* Willing and able to provide voluntary, written informed consent.

Exclusion Criteria:

* Acute illness within 2 weeks prior to dosing;
* History of any chronic illness or evidence of significant organic or psychiatric disease on medical history or physical examination which, in the opinion of the Investigator would confound the study results or present a risk to the subject;
* History of any clinically significant pulmonary conditions, within the last 2 years requiring admission to the hospital;
* Spirometry forced expiratory volume in one second (FEV1) and forced vital capacity (FVC) ratio less than 70%;
* If female, pregnant or lactating;
* Clinically significant illness or abnormality on physical examination, or ECG, including measure of the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle (QTc interval) >440 msec, on Screening or pre-dose 12-lead ECG;
* Resting heart rate while awake < 45 or > 90 b/m;
* Laboratory value(s) outside the laboratory reference range considered clinically significant (clinical chemistry, hematology, coagulation, ACTH, urinalysis, or pregnancy test).
* Presence of type I or type II diabetes;
* History of a severe allergic reaction to any drug or multiple food/drug allergies;
* Subjects with a formal diagnosis obstructive sleep apnea or having a score of >3 on the STOP-Bang questionnaire (see Appendix 4);
* Reported chronic (regular use for >1 month) use of medication of any kind (except contraceptives as described in the inclusion criteria), unless approved by the Sponsor;
* Reported use of any prescription drug within 14 days prior to dosing, any non-prescription drug or vitamin within 7 days prior to dosing, any known enzyme-inducer, enzyme-inhibitor, or other investigational drug within 30 days prior to dosing, or reported chronic exposure to enzyme-inducers such as paint solvents or pesticides within 30 days of dosing, unless approved by the Sponsor; hormonal contraceptive will be permitted if the subject has been using it for at least 12 weeks prior to dosing;
* History of alcohol or illicit drug abuse within the past two years, or current reported average alcohol intake > two alcoholic drinks per day (e.g., more than 24 oz. of beer, 10 oz. of wine, or 3 oz. of hard liquor);
* Regular use of tobacco or nicotine containing products within 1 year of study entry;
* Average consumption of ≥ 6 caffeine containing beverages per day;
* Consumption of alcohol within 72 hours prior to dosing, or a positive qualitative urine drug or cotinine screen, or positive oral screen for the presence of alcohol;
* Consumption of herbal supplements, grapefruit or grapefruit juice within 14 days before dosing;
* Blood donation of approximately 400 mL or more within 4 weeks or plasma donation within 2 weeks prior to dosing;
* Received an investigational product within 30 days of first dose in this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2013-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose (MTD) of single IV doses of AR09 | 4 hours
  Incidence of treatment-emergent adverse events (AE) by dose, including changes in temperature, respiratory rate, respiratory function at specified intervals post-dosing up to 24 hours.
  * Treatment-emergent changes in 12-lead electrocardiogram (ECG) recordings compared to pre-dose at specified intervals post-dosing and at Follow-Up including changes in heart rate and rhythm by dose at specified intervals post-dosing through 24 hours.
  * Treatment-emergent changes in group mean systolic and group mean diastolic blood pressure by dose at specified intervals post-dosing through 24 hours.
  * Treatment-emergent changes in clinical laboratory tests at specified intervals post-dosing and at Follow-Up.
  * Adrenocorticotropic hormone (ACTH) test to evaluate adrenal function pre and post dose.

SECONDARY OUTCOMES:
Characterize the single dose pharmacokinetics (PK) of IV doses of AR09 and its predominate metabolite, ADX892 | 24 hours
  Individual and group plasma concentration-time curves of AR09 and ADX892 (metabolite);
  * Individual and group maximum concentration (Cmax) and time to observed peak plasma concentration (Tmax);
  * For AR09, individual and group estimates of area under the curve (AUC) AUC 0-t, AUC 0-∞, terminal phase rate constant (λz), t1/2, systemic clearance (CL), and volumes of distribution (Vz and Vss).
  * For ADX892, individual and group estimates of AUC 0-t, AUC 0-∞, terminal phase rate constant (λz), and t1/2. Additional PK parameters for the metabolite, such as metabolite to parent ratios will be calculated on the basis of the available data.
  * Compartmental pharmacokinetic analysis may be employed depending upon the appearance of the AR09 and ADX892 plasma concentration-time profiles.

OTHER OUTCOMES:
Determine the safety and tolerability of single IV doses of AR09 | 24 hours
  Incidence of treatment-emergent adverse events (AE) by dose.
Identify doses of AR09 which produce moderate levels of sedation. | 4 hours
  * Mean Bispectral (BIS) index by dose at specified intervals post-dosing
  * Mean Modified Observer's Assessment of Alertness/Sedation (MOAA/S) score by dose at specified intervals post-dosing
  * Minute volume (tidal volume x respiratory rate)
  * End-tidal carbon dioxide (CO2) capnography by dose at specified intervals post-dosing
  * iPad-based cognitive tests by dose at specified intervals post-dosing

CONTACTS AND LOCATIONS:
Overall Officials: David MacLeod, MD, Principal Investigator — Duke University
Locations (1):
- Duke Clinical Research Unit, Durham, North Carolina, United States